CLINICAL TRIAL: NCT06992518
Title: The Effect of Bag Carrying Style on Gait Parameters in Healthy Adults: A Cross Sectional Study
Brief Title: The Effect of Bag Carrying Style on Gait Parameters in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gökçen Erol, MSc, PT, Istanbul University - Cerrahpasa
Other Study IDs: GErol2
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Gait Analysis; 3D Gait Analysis
Keywords: Posture; 3D Gait Analysis; Bag Carrying Styles; Healthy Adults

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational crossover study aims to evaluate how different bag carrying styles-backpack, shoulder bag, and handbag-may affect gait parameters in healthy adults. Fifteen participants will walk under four conditions (no bag and each of the three bag types with a load of 15% of body weight), with the order randomized. Gait will be assessed using a 3D motion capture system with integrated force plates. Posture and lower extremity muscle strength will also be evaluated for baseline characterization.

DETAILED DESCRIPTION:
This observational crossover study was conducted at a university-based Gait Analysis Center between October 2023 and October 2024, following ethical approval from the University Medical Research Ethics Committee (approval number: 2022-19/07, dated 09.12.2022). The study aimed to evaluate how different bag carrying styles-specifically, carrying a backpack, a shoulder bag, and a handbag-may influence gait parameters in healthy adults.

Fifteen volunteers aged 18 to 30 years who met predefined inclusion criteria were enrolled. Baseline posture was evaluated using the New York Posture Analysis (NYPA), and lower extremity muscle strength was assessed with a handheld myometer to ensure a consistent starting profile across participants. These values were recorded for characterization purposes only and were not analyzed in association with gait outcomes.

Each participant completed walking trials under four different conditions: walking without a bag, with a backpack, with a shoulder bag, and with a handbag. The order of these conditions was randomized for each participant. For each loaded condition, bags were adjusted to carry 15% of the individual's body weight. Participants walked barefoot at a self-selected pace on a 10-meter walkway while gait data were collected using a 3D motion analysis system (Vicon) integrated with force plates. Reflective markers were placed on anatomical reference points on the lower extremities.

Spatial-temporal, kinematic, and kinetic gait parameters were recorded in each condition, including stride length, cadence, joint angles, and joint power. Rest periods of at least three minutes were provided between walking conditions to reduce fatigue. All measurements were performed during a single session.

This study used a prospective crossover design in which each participant was observed under all four conditions. No therapeutic or clinical interventions were applied. The goal was to observe within-subject variability in gait characteristics associated with temporary exposure to different bag-carrying styles under standardized laboratory conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age,
* score above 45 on the New York Posture Analysis (NYPA)
* lower extremity muscle strength values measured with myometer greater than 24,
* No strenuous physical activity 48 hours before
* Being cooperative with the measurements and tests, and volunteering to participate in the study

Exclusion Criteria:

* Having a diagnosed orthopedic or neurological problem,
* Having visual problems,
* Having a body mass index of 30 kg/m² or more,
* Having pain complaints due to a history of trauma in the last 1 month,
* Having a leg length difference of more than 0.5 cm

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of 15 healthy volunteers who were selected using a simple random sampling method from among those who volunteered at Acıbadem Altunizade Hospital.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Kinetic Gait Parameters | Baseline
  Peak joint power values will be assessed using the Vicon 3D gait analysis system with integrated force plates. The following parameters will be recorded bilaterally under four bag-carrying conditions (no bag, backpack, shoulder bag, handbag):
  Maximum ankle power, maximum knee power, maximum hip power Unit of Measure: Watts per kilogram (W/kg)
Kinematic Gait Parameters | Baseline
  Joint angles will be calculated using 3D motion capture data for both right and left lower limbs during barefoot walking under four bag-carrying conditions (no bag, backpack, shoulder bag, handbag). The following maximum joint angles will be measured bilaterally:
  Ankle dorsiflexion, ankle plantarflexion, knee flexion, knee extension, hip flexion, hip extension, hip abduction, hip adduction, anterior pelvic tilt Unit of Measure: Degrees (°)
Spatiotemporal Gait Parameters | Baseline
  Spatiotemporal gait parameters will be measured using a 3D motion analysis system equipped with reflective markers and force platforms. The following variables will be assessed under four bag-carrying conditions (no bag, backpack, shoulder bag, handbag):
  Step length (meters), cadence (steps per minute), gait speed (meters per second), single support time (seconds), double support time (seconds) Each parameter will be recorded bilaterally where applicable. Values will be averaged from two selected trials per condition.
  Unit of Measure: Multiple (m, steps/min, s)

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız ANALAY AKBABA, Assoc. Prof, PT, Study Director — Istanbul University-Cerrahpasa,Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Division of Physiotherapy and Rehabilitation
Locations (1):
- Istanbul University - Cerrahpasa, Faculty of Health Sciences, Büyükçekmece Campus, Alkent 2000 Mah. Yiğittürk Street No:5/9/1, Büyükçekmece/Istanbul, Turkey, Istanbul, büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers

REFERENCES:
- [Background] Ozgul B, Akalan NE, Kuchimov S, Uygur F, Temelli Y, Polat MG. Effects of unilateral backpack carriage on biomechanics of gait in adolescents: a kinematic analysis. Acta Orthop Traumatol Turc. 2012;46(4):269-74. doi: 10.3944/aott.2012.2678. PMID 22951758
- [Background] Cottalorda J, Rahmani A, Diop M, Gautheron V, Ebermeyer E, Belli A. Influence of school bag carrying on gait kinetics. J Pediatr Orthop B. 2003 Nov;12(6):357-64. doi: 10.1097/01.bpb.0000078270.58527.1f. PMID 14530691
- [Background] Connolly BH, Cook B, Hunter S, Laughter M, Mills A, Nordtvedt N, Bush A. Effects of backpack carriage on gait parameters in children. Pediatr Phys Ther. 2008 Winter;20(4):347-55. doi: 10.1097/PEP.0b013e31818a0f8f. PMID 19011525
- [Background] Alamoudi, M., Travascio, F., Onar-Thomas, A., Eltoukhy, M., & Asfour, S. (2018). The effects of different carrying methods on locomotion stability, gait spatio-temporal parameters and spinal stresses. International Journal of Industrial Ergonomics, 67, 81-88.
- [Background] Ahn, J. (2006). The effects of asymmetric load of shoulder bag on trunk and pelvis movement patterns of normal adult during gait. The Graduate School of Health and Environment Yonsei University, Master's thesis.
- [Background] Abaraogu UO, Ugwa WO, Onwuka E, Orji E. Effect of single and double backpack strap loading on gait and perceived exertion of young adults. J Back Musculoskelet Rehabil. 2016;29(1):109-15. doi: 10.3233/BMR-150605. PMID 26406186